CLINICAL TRIAL: NCT00319618
Title: A Randomised Phase II Study: Treatment With Daily p.o. Iressa™ (ZD1839) or Placebo in Combination With Weekly IV Infusion of Docetaxel in Patients With Metastatic Breast Cancer
Brief Title: Combination Weekly Taxotere™ With Iressa™ /Placebo in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0128
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Docetaxel

INTERVENTIONS:
Drug: Gefitinib
Drug: Docetaxel

SUMMARY:
The purpose of this study is to determine if combination therapy of weekly Taxotere™ with Iressa™ will increase the objective responses in measurable leasions in metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mammary carcinoma

Exclusion Criteria:

* prior taxane chemotherapy for metastatic disease or prior treatment with tyrosine kinase inhibitors inhibiting the EGF receptor.
* Prior hormone treatment or one type of anthracycline based treatment regimen without taxane for metastatic disease is allowed prior to inclusion.
* If the patient has been treated in the adjuvant or neoadjuvant setting with taxanes, inclusion is allowed when the first cycle of trial medication is started 12 months after the last course of adjuvant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2003-06; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Objective tumour response (CR + PR) per RECIST criteria

SECONDARY OUTCOMES:
Time to progression and response duration
Exploratory outcomes: Objective tumour response in relation to ER, PgR, erb-B1 and erb-B2 receptor status and reduction in the number of malignant cells present in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Norway Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Oslo, Norway